CLINICAL TRIAL: NCT05483348
Title: Clinical Predictive Factors of Success of Hysteroscopic Endometrial Ablation/Resection; Retrospective Study at a Tertiary University Hospital
Brief Title: Clinical Predictive Factors of Success of Hysteroscopic Endometrial Ablation/Resection
Status: Completed | Type: Observational
Sponsor: Naser Al-Husban (Other)
Responsible Party: Sponsor-Investigator, Naser Al-Husban, Assistant professor of obstetrics and gynecology, the university of jordan, University of Jordan
Organization: University of Jordan (Other)
Other Study IDs: 4276
Record Dates: First submitted 2022-07-16; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Uterine Bleeding; Treatment Failures; Prognostic Factors
Keywords: Endometrial Ablation Technique; Uterine Bleeding; Treatment Failures; Prognostic Factors
MeSH Terms: conditions — Uterine Hemorrhage | interventions — Endometrial Ablation Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients who had successful endometrial ablation: Patients included in this group experienced abnormal uterine bleeding and underwent endometrial ablation. Successful ablation was defined as not undergoing subsequent gynecological procedures such as hysterectomy for any benign indication, D&C or repeat ablation within 36 months after the endometrial ablation.
  Interventions: Procedure: Endometrial Ablation
- Patients who had unsuccessful endometrial ablation: Patients included in this group experienced abnormal uterine bleeding and underwent endometrial ablation. Unsuccessful ablation was defined as undergoing subsequent gynecological procedures such as hysterectomy for any benign indication, D&C or repeat ablation within 36 months after the endometrial ablation.
  Interventions: Procedure: Endometrial Ablation; Procedure: Repeated gynecological procedure

INTERVENTIONS:
Procedure: Endometrial Ablation — Thermal endometrial ablation
Procedure: Repeated gynecological procedure — subsequent gynecological procedures such as hysterectomy for any benign indication, D&C or repeat ablation.
  Groups: Patients who had unsuccessful endometrial ablation

SUMMARY:
To determine the predictive factors of endometrial ablation failure in the management of uterine bleeding.

DETAILED DESCRIPTION:
This is a retrospective cohort study for women who have been treated with Thermal endometrial ablation due to uterine bleeding. The main purpose of this study is to demonstrate the possible risk factors associated with endometrial ablation failure causing patients to need subsequent gynecological procedures or undergoing hysterectomy for definitive treatment. Such efforts are made in order to anticipate the morbidity and mortality associated with patients in such conditions and to effectively stratify those patients to appropriate treatment techniques.

ELIGIBILITY:
Inclusion Criteria:

* All patients who had their endometrial ablation at Jordan University Hospital.

Exclusion Criteria:

* Patients whose index ablation or subsequent re-intervention could not be confirmed in detailed operative reports were excluded

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who had attended the gynecology department at Jordan University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Clinical Predictive factors of successful endometrial ablation | from September 2016 through February 2022
  the outcome of hysteroscopic endometrial ablation whether it was a failure or a success; failure was defined as persistent of heavy bleeding after the ablation.

SECONDARY OUTCOMES:
The failure rate of endometrial ablation for uterine bleeding | from September 2016 through February 2022
  To find the failure rate of endometrial ablation that is done for uterine bleeding
Subsequent gynecological procedures after failed ablation | from September 2016 through February 2022
  To find the subsequent gynecological procedures that patients with unsuccessful ablation had

CONTACTS AND LOCATIONS:
Overall Officials: Naser AL- Husban, MD, Principal Investigator — Assistant professor of obstetrics and gynecology, the university of jordan
Locations (1):
- Jordan University Hospital, Amman, Al Jubaiha, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available

REFERENCES:
- [Result] Wortman M. Late-onset endometrial ablation failure. Case Rep Womens Health. 2017 Jul 12;15:11-28. doi: 10.1016/j.crwh.2017.07.001. eCollection 2017 Jul. PMID 29593995
- [Result] Riley KA, Davies MF, Harkins GJ. Characteristics of patients undergoing hysterectomy for failed endometrial ablation. JSLS. 2013 Oct-Dec;17(4):503-7. doi: 10.4293/108680813X13693422520602. PMID 24398189
- [Result] Smithling KR, Savella G, Raker CA, Matteson KA. Preoperative uterine bleeding pattern and risk of endometrial ablation failure. Am J Obstet Gynecol. 2014 Nov;211(5):556.e1-6. doi: 10.1016/j.ajog.2014.07.005. Epub 2014 Jul 11. PMID 25019488
- [Result] El-Nashar SA, Hopkins MR, Creedon DJ, St Sauver JL, Weaver AL, McGree ME, Cliby WA, Famuyide AO. Prediction of treatment outcomes after global endometrial ablation. Obstet Gynecol. 2009 Jan;113(1):97-106. doi: 10.1097/AOG.0b013e31818f5a8d. PMID 19104365
- [Result] Gemer O, Kruchkovich J, Huerta M, Kapustian V, Kroll D, Anteby E. Perioperative predictors of successful hysteroscopic endometrial ablation. Gynecol Obstet Invest. 2007;63(4):205-8. doi: 10.1159/000097847. Epub 2006 Dec 7. PMID 17159353
- [Result] Shazly SA, Famuyide AO, El-Nashar SA, Breitkopf DM, Hopkins MR, Laughlin-Tommaso SK. Intraoperative Predictors of Long-term Outcomes After Radiofrequency Endometrial Ablation. J Minim Invasive Gynecol. 2016 May-Jun;23(4):582-9. doi: 10.1016/j.jmig.2016.02.002. Epub 2016 Feb 9. PMID 26867699